CLINICAL TRIAL: NCT00125281
Title: S-Adenosyl Methionine for Symptomatic Treatment of Primary Biliary Cirrhosis
Brief Title: SAMe to Treat Biliary Cirrhosis Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jay H. Hoofnagle, M.D./National Institute of Diabetes and Digestive and Kidney Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 050207; 05-DK-0207
Record Dates: First submitted 2005-07-29; First posted 2005-07-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-02

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: Fatigue; Cirrhosis; S-Adenosyl Methionine; Primary Biliary Cirrhosis; Pruritus; Symptomatic Releif; Serum Liver-Related Enzymes; PBC; Liver Disease
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fatigue; Fibrosis; Pruritus; Liver Diseases | interventions — S-Adenosylmethionine; Capsules

INTERVENTIONS:
Drug: S-adenosyl-methionine (SAMe) capsules

SUMMARY:
This study will examine the effect of S-adenosyl methionine (SAMe) on itching and fatigue in patients with primary biliary cirrhosis, a disease of the small bile ducts in the liver. Ursodiol, the only currently available treatment for biliary cirrhosis, does not cure the disease, and many people continue to have symptoms or liver test abnormalities despite treatment. SAMe is a naturally occurring substance found in most cells of the body. The highest levels of the substance are produced by the liver, where it helps to rid the body of toxins and breakdown products of metabolism. Studies in Europe suggest that SAMe may help to: 1) decrease the fatigue and itching that are common in persons with liver problems, and 2) decrease levels of liver enzymes in the blood, suggesting that it may decrease the amount of liver injury.

Patients 21 years of age or older with primary biliary cirrhosis who are taking ursodiol and have symptoms of itching or fatigue may be eligible for this study. Candidates are screened with a medical history, physical examination, review of medical records, routine blood tests, and a symptoms rating scale.

Participants stop all medications for itching 4 weeks before starting the study, but continue to take ursodiol during the 42-week trial. On entering the study, patients are assigned to take either SAMe or placebo tablets twice a day for 12 weeks. While taking the medications, they are followed in the clinic every 2 weeks for the first month and then every 4 weeks to fill out symptoms questionnaires and have a short medical evaluation and blood tests. At the end of 12 weeks, treatment is interrupted for a 2-week "wash-out" period, after which patients begin a 12-week crossover treatment; that is, patients who were taking SAMe are switched to placebo, and those who were taking placebo are switched to SAMe.

After completing the second 12-week treatment course, patients come to the clinic at 4, 8, and 12 weeks to fill out symptoms questionnaires and have a medical evaluation and blood tests. At the last visit, patients are told which type of tablet they received during the two courses of treatment. SAMe is available without prescription in many forms as an over-the-counter medication.

DETAILED DESCRIPTION:
To assess the efficacy of S-adenosyl methionine (SAMe) in symptomatic relief of primary biliary cirrhosis (PBC), we will treat up to 50 patients with either SAM-e (800 mg BID) or placebo for 12 weeks in a cross-over, double-blind placebo-controlled study.

S-adenosyl methionine is a nutritional supplement which is available as an over-the-counter formula and is used for treatment of depression and arthritic pain. SAMe is produced in virtually all cells and participates in many biochemical pathways as a major methyl contributor. Intracellular levels of SAMe are often decreased in advanced liver disease. At present SAMe is undergoing extensive evaluation in a large multicenter, randomized controlled trial as an adjunctive therapy of alcoholic liver disease. SAMe has also been evaluated in patients with intrahepatic cholestasis and cholestasis of pregnancy with promising effects of relieving pruritus and fatigue and improving serum liver associated enzymes.

In this study, we will recruit patients with PBC who have pruritus or fatigue despite therapy with ursodiol (the currently recommended therapy of PBC which is partially effective in relieving pruritus and fatigue). After medical evaluation and a brief period of monitoring, patients will be randomized to receive either SAMe or placebo given in oral form in similar appearing capsules twice daily. Patients will be followed at regular intervals for symptoms as monitored by validated questionnaires as well as for side effects and serum biochemical and hematological tests. After 12 weeks, therapy will be withdrawn for 2 weeks and patients will then be switched to the alternative capsules, either SAMe or placebo, for another 12 weeks. The primary endpoints of therapy will be improvements in symptoms of pruritus or fatigue or both. Secondary endpoints will be improvements in serum biochemical liver related enzymes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age at entry at least 21 years old.

Pathologically diagnosed primary biliary cirrhosis (made by a liver biopsy performed within 10 years of enrollment) with receipt of stable doses of ursodiol for at least 6 months before enrollment. The dose of urosodiol will be adjusted to achieve stable serum liver enzymes levels.

Symptoms of itching or fatigue or both. The presence of symptoms will be verified by medical history, symptom questionnaire and visual analogue scales (results greater than 20 mm) on at least two screening visits.

Written informed consent.

EXCLUSION CRITERIA:

Evidence of another form of liver disease.

Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg) in serum.

Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA in serum.

Primary sclerosing cholangitis as defined by liver histology.

Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.

Autoimmune hepatitis as defined by antinuclear antibody (ANA) of 3 EU or greater (ELISA) and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy for autoimmune hepatitis.

Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.

Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D. Patients with iron saturation indices of greater than 45% and serum ferritin levels of greater than 300 ng/ml for men and greater than or equal to 250 ng/ml for women will undergo genetic testing for C282Y and H63D.

Drug induced liver disease as defined on the basis of typical exposure and history.

Bile duct obstruction as suggested by imaging studies done within the previous six months.

Decompensated liver disease as defined by a Child-Pugh score of 7 or greater.

Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease with hypoxia, renal failure, organ transplantation, serious psychiatric disease including depression, malignancy and any other conditions that in the opinion of the investigator would preclude treatment. Patients who are suffering from severe depression defined by a score of greater than or equal to 25 in CES-D screening test will not be eligible for enrollment.

Known HIV infection.

Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.

Pregnancy, lactation or inability to practice adequate contraception in women in child bearing age.

Evidence of hepatocellular carcinoma as shown by a liver mass on imaging studies or alphafetoprotein levels greater than 200 ng/ml.

Any other condition, which in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study.

History of hypersensitivity reactions to S-adenosyl methionine.

Serum creatinine greater than 1.5mg/dl in men and greater than 1.4 mg/dl for women.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-07-25; Primary Completion 2007-07-31 (Actual); Study Completion 2008-07-02 (Actual)

PRIMARY OUTCOMES:
Improvement in symptoms as assessed by validated questionnaires and visual analogue scales administered at 2 to 4 week intervals during therapy. | 12 weeks of therapy

SECONDARY OUTCOMES:
Improvement in serum alanine aminotransferase and alkaline phosphatase. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] LLOYD-THOMAS HG, SHERLOCK S. Testosterone therapy for the pruritus of obstructive jaundice. Br Med J. 1952 Dec 13;2(4797):1289-91. doi: 10.1136/bmj.2.4797.1289. No abstract available. PMID 12997743